CLINICAL TRIAL: NCT01750307
Title: The Relationship of Essential Fatty Acids to Cognitive Electrophysiological and Behavioural Function in Adults With Attention Deficit Hyperactivity Disorder and Controls
Brief Title: The Relationship of Essential Fatty Acids to Adult ADHD: The OCEAN Study (Oils and Cognitive Effects in Adult ADHD Neurodevelopment)
Acronym: OCEAN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Responsible Party: Principal Investigator, Philip Asherson, Professor, King's College London
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OCEAN protocol
Record Dates: First submitted 2012-12-12; First posted 2012-12-17 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-12

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
Keywords: Attention Deficit Hyperactivity Disorder (ADHD); Essential fatty acids (EFAs); Electroencephalography (EEG); Event-related potential (ERP); Omega 3; Randomised Control Trial; Fish oil; Supplementation; Reading; Spelling; Behaviour; Emotional lability
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fatty acid supplementation (Experimental): 4 capsules to be taken daily
  Interventions: Dietary Supplement: Experimental fatty acid supplementation
- Medium Chain Triglyceride (MCT) oil softgel (Placebo Comparator): 4 capsules to be taken daily
  Interventions: Dietary Supplement: Placebo comparator: MCT oil softgel

INTERVENTIONS:
Dietary Supplement: Experimental fatty acid supplementation — 4 x capsules per day. Daily dose: 1584mg EFA
  Other Names: Essential fatty acid: Eye Q triple (product code: FO-5274ART)
  Arms: Fatty acid supplementation
Dietary Supplement: Placebo comparator: MCT oil softgel — 4 x capsules per day. Medium chain triglyceride pill manufactured to mimic essential fatty acid pill
  Other Names: MCT oil softgel (Product code: GL-5200ART)
  Arms: Medium Chain Triglyceride (MCT) oil softgel

SUMMARY:
Brief summary

The aim of the study is to provide preliminary data on the relationship of Essential Fatty Acids (EFAs) to cognitive and electrophysiological measures of brain and behavioural functions in adults with attention deficit hyperactivity disorder (ADHD) and controls. This main aim will be achieved in two ways. First the investigators will measure the relationship of the various measures to blood levels of EFAs in ADHD cases and controls. Secondly, the potential effects of dietary supplementation with EFAs on cognitive-electrophysiological and behavioural measures in ADHD cases will be investigated. We will evaluate the extent to which changes in neuronal activity and cognitive performance are related to behavioural and functional measures over time. This is to be carried out by conducting a randomised controlled trial of fish oil supplementation in adults with ADHD (The OCEAN study: Oils and Cognitive Effects in Adult Neurodevelopment).

The study design will be a 6-month double blind placebo control study with a group of 80 adults with a diagnosis of ADHD. The group will be divided into 40 participants who receive EFA dietary supplements and 40 who receive placebo, over a 6-month period. Allocation to EFA dietary supplementation and placebo groups will be randomly allocated and blind to both the investigator and participants. In addition a sample of 30 controls will take part in baseline levels of assessment and be used for case-control comparisons to investigate the links between EFA blood levels and cognitive-electrophysiological function at one time point.

The study design will enable preliminary data to address the following hypotheses:

1. Changes in cognitive and electrophysiological function (neuronal activity) will be found following supplementation with dietary EFAs.
2. Changes in cognition and/or brain activity will be related to blood levels of EFAs.
3. Changes in cognitive performance and electrophysiological parameters will correlate with behavioural function, affective regulation or functional impairments.
4. At baseline, case-control differences in EFA blood-levels will be found which will be linked to cognitive and electrophysiological function.

ELIGIBILITY:
Inclusion Criteria:

* Cases:
* Clinical diagnosis of ADHD (combined or inattentive type)
* Controls:
* Screen below threshold for ADHD

Exclusion Criteria:

* Cases:
* Autism spectrum disorder
* Recurrent major depression
* Bipolar I disorder
* Psychotic disorders
* Obsessive compulsive disorder
* Learning difficulties (IQ < 80)
* Neurological problems
* Drug abuse
* Those who are already taking EFA supplements
* Metabolic conditions
* Infectious diseases
* Controls:
* ADHD
* All other exclusion criteria for cases as above

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-09; Primary Completion 2014-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
The relationship of essential fatty acids to cognitive and electrophysiological measures of brain and behavioural function | 6 months
  Brain function will be measured using direct current (DC) electroencephalography (EEG) in participants first while they are at rest and second during 4 cognitive tasks. Behavioural function will be measured through assessment of reading and spelling, emotional lability, ADHD symptoms and other self-ratings of behaviour (such as executive function). These measures will be related to the effect of dietary supplementation and blood levels of EFAs in adults with ADHD.

SECONDARY OUTCOMES:
The relationship of essential fatty acids to ADHD | 0 months
  This will be assessed by recording blood levels of EFAs in cases and controls at baseline assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Asherson, Principal Investigator — King's College London
Locations (1):
- Social, genetic and developmental psychiatry, Institute of Psychiatry, King's College London, London, London, United Kingdom